CLINICAL TRIAL: NCT02295748
Title: An Open-Label, Multi-Center, Long-Term Extension Study to Evaluate the Safety and Tolerability of Orally Administrated Deflazacort in Children and Adolescent Subjects With Duchenne Muscular Dystrophy
Brief Title: An Open-Label, Long-Term Extension Study to Evaluate the Safety and Tolerability Deflazacort
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-104-CL-022OLE
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-01

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — deflazacort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deflazacort (Experimental): 0.9 mg/kg oral deflazacort (between 2 to 12 x 6mg tablets based on body weight) will be administered daily.
  Interventions: Drug: Deflazacort

INTERVENTIONS:
Drug: Deflazacort — Deflazacort, a glucocorticoid with anti-inflammatory and immunosuppressive effects, is used in treating a variety of diseases. Pharmacologically it is an inactive pro-drug which is metabolized rapidly to the active drug 21-desacetyldeflazacort.
  Other Names: DFZ

SUMMARY:
This is an open label, long-term extension study in approximately 24 male DMD subjects consisting of children (ages 4-12, inclusive) and adolescents (ages 13-16, inclusive) who participated in the MP-104-CL-005 PK study.

DETAILED DESCRIPTION:
This is an open label, long-term extension study in approximately 24 male DMD subjects consisting of children (ages 4-12, inclusive) and adolescents (ages 13-16, inclusive) who participated in the MP-104-CL-005 PK study.

Subjects may have received up to 8 (+2 days) doses of deflazacort during the MP-104-CL-005 PK study, at which point treatment will be continued at the same dose and frequency until such time that deflazacort becomes commercially available or the study is terminated. Concomitant corticosteroid therapy will be prohibited during the study while the subject is taking deflazacort.

Subjects will be given medication to take at home for once-daily, morning dosing following the 8 hour PK sample on Day 8 (+2 days) of the MP-104-CL-005 PK study. Subjects will begin dosing at home the day following Day 8 (+2 days) of the MP-104-CL-005 PK study.

Safety will be monitored throughout the study by repeated clinical and laboratory evaluations every 3 months for the first year, and then every 3 or 6 months, depending on subjects' disease status.

Subjects will be contacted via telephone between study visits to determine if any adverse events (AE) have occurred since the last study visit. Subjects who terminate the study early will be contacted if the Principal Investigator (PI) deems necessary.

Treatment will be continued for a maximum of three years or until such time that deflazacort becomes commercially available or the study is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is capable of understanding and complying with protocol requirements.
* Subject or, when applicable, the subject's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* If above the age of 7, the subject signs and dates a written, informed assent form (IAF) and any required privacy authorization prior to the initiation of any study procedures. Subjects under age 7 at the time of study entry who turn age 7 will sign and date a written informed assent form (IAF) at the visit following their 7th birthday, if required by the site's IRB.
* Subject participated in and received at least one dose of study medication in the MP-104-CL-005 protocol.
* The subject must have confirmed diagnosis of Duchenne Muscular Dystrophy defined as:

  1. onset of weakness before 5 years of age;
  2. proximal muscle weakness;
  3. increased serum creatine kinase more than 10 times the upper limit of normal (ULN);
  4. muscle biopsy and dystrophin analyses consistent with DMD or DNA mutation and analysis by PCR or Southern blot techniques to detect gene deletions.
* The subject weighs at least 13 kg and has a body mass index (BMI) of ≤ 40 kg/m2.
* Willingness and ability to comply with scheduled visits, oral drug administration, and study procedures including blood sample draws for safety labs.
* Up to date on all childhood vaccinations, including varicella vaccine (chicken pox).
* Baseline health is judged to be stable based on medical history, physical examination, laboratory profiles, vital signs, or ECGs at screening, as deemed by the Investigator.
* Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dose.
* The subject is able to take tablets.

Exclusion Criteria:

* The subject has received any investigational compound and/or has participated in another clinical study within 90 days prior to study treatment with the exception of MP-104-CL-005, observational cohort studies or non-interventional studies.
* The subject is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g. spouse, parent, child, sibling) or may consent under duress.
* Any significant finding on the Columbia suicide severity rating scale (C SSRS) for subjects (ages 12-16, inclusive), in the opinion of the PI, warrants exclusion from this study.
* The subject has, in the judgment of the, clinically significant abnormal clinical chemistry laboratory parameters that may affect safety at Day 0.
* The subject has, in the judgment of the Investigator, a history or current medical condition that could affect safety including, but not limited to:

  1. Major renal or hepatic impairment
  2. Immunosuppression or other contraindications for corticosteroid treatment
  3. History of chronic systemic fungal or viral infections
  4. Diabetes mellitus
  5. Idiopathic hypocalciuria
  6. Symptomatic cardiomyopathy at Day 0
* The subject has a history of hypersensitivity or allergic reaction to steroids or their formulations including, but not limited to lactose, sucrose, etc.
* Inability to take tablets as assessed by site investigator.
* Subject is mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected during the conduct of the study.
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* Positive urine drug or alcohol results at Day 0.
* Hemoglobin level below the lower limit of normal at Day 0.

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Number, frequency, and severity of adverse events | 3 years
  Long-term safety and tolerability will be characterized by the number, frequency, and severity of adverse events from Day 1 through End of Study or Early Termination.

CONTACTS AND LOCATIONS:
Overall Officials: Marathon Bioscience Center, Study Director — Marathon Pharmaceuticals
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Rochester, Rochester, New York
  - University of Utah, Salt Lake City, Utah